CLINICAL TRIAL: NCT01933178
Title: Inter and Intra Examiner Reproducibility of Anterior Segment Optical Coherence Tomography (AS-OCT) for Imaging Conjunctivochalasis
Brief Title: Reproducibility of Anterior Segment Optical Coherence Tomography (AS-OCT) for Imaging Conjunctivochalasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Louis Tong, Clinician-Scientist, Senior Consultant, Singapore National Eye Centre
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: R1029/44/2013; 2013/328/A (Other: SingHealth Centralised Institutional Review Board)
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Dry Eyes
Keywords: Dry eyes; Cirrus AS-OCT; Excess folds of the conjunctiva
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cirrus AS-OCT (Other)
  Interventions: Device: Cirrus AS-OCT

INTERVENTIONS:
Device: Cirrus AS-OCT

SUMMARY:
Conjunctivochalasis refers to loose redundant, non-edematous inferior conjunctiva that is situated between the globe and lower eyelid, and usually it occurs bilaterally. It has been reported to cause ocular discomfort, tear instability, alteration of tear spreading and subsequently dry eye, which is a common condition that affects vision and quality of life in patients. This condition has also been reported to be associated with aging and ocular surface inflammation.

The assessment of conjunctivochalasis was traditionally based on silt lamp examination and this may be cumbersome and highly subjective. Only recently, researchers have advocated the use of imaging and more objective documentation by anterior segment optical coherence tomography (AS-OCT), using Fourier-Domain RTVue-100 OCT. The AS-OCT is an imaging method that documents the tear meniscus and prolapse of conjunctiva into the tear meniscus in a safe, rapid and non-invasive way. Image analysis on the area of prolapsed conjunctiva can then be used to ascertain the severity of conjunctivochalasis. We propose the use of HD-Cirrus AS-OCT for the imaging of conjunctivochalasis, since this technique provides more magnified and colored digital images, which helps to delineate different tissues and serves as a better education tool for patients.

This current study aims to investigative the inter and intra examiner reproducibility of imaging conjunctivochalasis using HD-Cirrus AS-OCT, using patients from the dry eye clinic from the Singapore National Eye Centre. These patients will be asked to come to the centre for imaging and have three scans of the same eye performed in one session by two trained investigators consecutively. The resulting limits of repeatability will be very useful for us to follow up patients who undergo surgical or diathermy treatment for conjunctivochalasis, and for sample size calculation in the planning of interventional studies.

DETAILED DESCRIPTION:
This study will be conducted in compliance with the protocol, SGCP and the applicable regulatory requirements.

Dry eye is a condition that affects 5-35% of the population9. Common symptoms of this condition include eye irritation, heaviness of the eyelids, visual disturbances, tearing and light sensitivity9-11. This significantly impacts the quality of life and vision of dry eye patients. In addition, there is a significant socio-economic burden. In 2009, 54,051 patients sought treatment for dry eye in the Singapore National Eye Centre (SNEC). In total, the costs for dry eye medication amounted to $181,354.1712. Additionally, dry eye affects work productivity which further adds on to the socio-economic burden9,12.

Currently, the diagnosis and assessment of dry eye is hindered by tests that have poor repeatability, some of which cause discomfort due to their invasiveness. As a result most clinical studies involving dry eye treatment rely on symptomatic improvements as a primary outcome measure. However, symptomatic improvements are a poor measure in determining treatment effectiveness. This may be a result of disease progression that damages nerves which consequently desensitizes the eye. Also, it is not uncommon that patients feel a reduction of discomfort of the eye before objective improvements can be noted by the clinician. An assessment based on symptoms alone is therefore inappropriate11.

Over the last few years, SNEC/SERI has built up a dedicated team of dry eye researchers for trials and evaluation of diagnostic devices. There is an increasing interest internationally, especially from industry, to partner us for testing of commercial products.

The anterior segment optical coherence tomography (AS-OCT) is an imaging device that allows clinicians to acquire images of the conjunctivochalasis in a safe and non-invasive manner. The device utilizes infra-red light which is reflected on the eye surface. The reflection, affected by the thickness of the tissue, is then used to generate an image. It also was found to correlate with other less repeatable diagnostic tests, such as tear film break-up time (TBUT), which measures tear film stability.

The applicability of the HD-Cirrus AS-OCT in dry eye research has not been extensively tested. It is also not known if HD-Cirrus AS-OCT would be able to image repeatable and reproducible results. It is highly cost effective for the study team here to evaluate the HD-Cirrus ASOCT because it is already available in the trial center, being purchased from other grant funding.

Figure 1 illustrates the high magnification coloured images taken from our preliminary study of normal tear meniscus and conjunctivochalasis using the HD-Cirrus AS-OCT.

Figure 1: Cirrus AS-OCT images of normal tear meniscus and conjunctivochalasis

Clinical importance Should this modality of imaging be validated or shown to be reproducible, it can then be incorporated into our protocol/workflow for assessment and monitoring of dry eye treatment in our centre and will greatly enhance our capability to perform clinical trials and increase our international reputation.

Study Objectives and Purpose The primary purpose is to evaluate inter and intra examiner repeatability of the HD-Cirrus AS-OCT imaging system to capture conjunctivochalasis.

Study design:

Prospective study

Rationale:

Repeatability is an important issue in the objective assessment of dry eye. There is lack of studies that investigate the HD-Cirrus AS-OCT for assessment of conjunctivochalasis. The HD-Cirrus AS-OCT is potentially useful as a non-invasive procedure for objective measurements of the conjunctivochalasis.

Methods:

Participants and target sample size 10 patients with symptomatic dry eye and clinically suspected conjunctivochalasis (presence of lid parallel conjunctival folds) from Singapore National Eye Centre will be recruited for this study. 10 healthy volunteers with no symptoms of dry eyes will be recruited for this study as controls. Each volunteer will also be given a study serial number to ensure anonymity.

All 20 volunteers will participate in the AS-OCT study.

Visit schedules One visit is required for paticipants.

Duration of study:

8 months.

Procedures:

Participants will need to stay for the study for 60 minutes.

1. Assessment of Dry Eye Symptoms Basic biodata such as age, race, gender will be recorded. Participants' habitual visual acuity will also be documented. Participants will be asked to score and fill up a dry eye questionnaire that assesses the symptomatic severity of dry eyes and the extent of its disruption to daily activities.
2. HD-Cirrus AS-OCT for the assessment of proplasped conjunctiva Participants are randomly assigned to first examiner, followed by the second examiner. Each examiner will capture 2 sets of scans from the randomly chosen eye of the participants.

   During the acquisition, the participants place their chins on a chin rest and look at a fixation light/target. This whole procedure of should take about 10 minutes. The participants are allowed to blink freely except for during the acquisition time of less than 5 seconds.

   The eye is scanned at 3 vertical positions: inferior temporal (IT), inferior central (IC) and inferior nasal (IN), as shown in figure 2. In milder case of conjunctivochalasis, the prolapse of conjunctiva into the tear menicus is more prominent in the IT scan than IC scan. Therefore, it is important to obtain prolapsed conjunctiva at different region of the tear meniscus.

   Figure 2: Imaging prolapsed conjunctiva at different region of the tear meniscus
3. Fluorescein Dye Tear Break-up Time (TBUT) Fluorescein dye is introduced onto the lower eyelid by a wetted fluorescein strip. The tear film will then be observed with blue light using a slit lamp to the point where it breaks. The time from the previous blink to the breaking of the tear film will be recorded to the nearest second.
4. Fluorescein Dye Corneal Staining After fluorescein dye is introduced, the cornea will be examined for green stains indicating epithelial erosion, a sign of damage due to dryness. The number of green stains and their ocation on the cornea (superior, central, inferior, temporal, nasal fields) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers that are medically fit and willing to participate in this study.

Exclusion Criteria:

* No eye surgery done within the previous 3 months
* Active ocular infection or pterygium that may affect tear film stability.
* Any other specified reason as determined by clinical investigator.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The repeatabilty of objective conjunctivochalasis measurements of HD-Cirrus AS-OCT from the same examiner, and between the two examiners | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Louis Tong, PhD, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore, Singapore